CLINICAL TRIAL: NCT01014338
Title: ACE-inhibition and Mechanisms of Skeletal Muscle Weakness in Chronic Obstructive Pulmonary Disease
Brief Title: Angiotensin-converting Enzyme (ACE)-Inhibition and Mechanisms of Skeletal Muscle Weakness in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P15099; ISRCTN05581879 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fosinopril; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE-inhibitor (Active Comparator)
  Interventions: Drug: Fosinopril
- Sugar Pill (Placebo Comparator)
  Interventions: Other: lactose

INTERVENTIONS:
Drug: Fosinopril — 10mg od
  Arms: ACE-inhibitor
Other: lactose — placebo
  Arms: Sugar Pill

SUMMARY:
A double blind randomised placebo controlled parallel trial of the effect of fosinopril, an angiotensin converting enzyme inhibitor, on the quadriceps muscle in 80 COPD patients who have quadriceps weakness. Patients will have a baseline assessment including measures of quadriceps strength and endurance and a quadriceps biopsy. Patients with weakness will be randomised to ACE inhibitor or placebo and re-assessed after three months of treatment.

The investigators aim to show that ACE-inhibition will alter the IGF-1/AKT/FoXO/atrogene pathways involved in muscle wasting in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with COPD diagnosed according to GOLD criteria.

Exclusion Criteria:

* Clinically unstable patients (within one month of exacerbation), those with a permanent pacemaker (which is a contraindication to magnetic stimulation), or significant co-morbidity, patients with an accepted indication for ACE inhibition (left ventricular dysfunction, diabetes) or a contraindication such as renovascular disease; creatinine clearance (estimated) <50); hypotension; use of anticoagulants (contra-indication to biopsy) or ACE-I or ATII receptor antagonists.
* Allergy to ACE-inhibitors.
* Pregnancy.

Patients will not be enrolled within three months of participation in a pulmonary rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes in phosphorylation of components of the atrogene pathway | 3 months

SECONDARY OUTCOMES:
Quadriceps endurance assessed non-volitionally | 3 months
Effect of ACE-I on quadriceps maximum voluntary contraction force | 3 months
Effect of ACE-I on quadriceps bulk (cross-sectional area) | 3 months
Effect of ACE-I on systemic inflammation and serum IGF-1 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hopkinson, MRCP, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Background] Hopkinson NS, Nickol AH, Payne J, Hawe E, Man WD, Moxham J, Montgomery H, Polkey MI. Angiotensin converting enzyme genotype and strength in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Aug 15;170(4):395-9. doi: 10.1164/rccm.200304-578OC. Epub 2004 Apr 29. PMID 15117739
- [Background] Swallow EB, Reyes D, Hopkinson NS, Man WD, Porcher R, Cetti EJ, Moore AJ, Moxham J, Polkey MI. Quadriceps strength predicts mortality in patients with moderate to severe chronic obstructive pulmonary disease. Thorax. 2007 Feb;62(2):115-20. doi: 10.1136/thx.2006.062026. Epub 2006 Nov 7. PMID 17090575
- [Background] Hopkinson NS, Eleftheriou KI, Payne J, Nickol AH, Hawe E, Moxham J, Montgomery H, Polkey MI. +9/+9 Homozygosity of the bradykinin receptor gene polymorphism is associated with reduced fat-free mass in chronic obstructive pulmonary disease. Am J Clin Nutr. 2006 Apr;83(4):912-7. doi: 10.1093/ajcn/83.4.912. PMID 16600946
- [Background] Andreas S, Herrmann-Lingen C, Raupach T, Luthje L, Fabricius JA, Hruska N, Korber W, Buchner B, Criee CP, Hasenfuss G, Calverley P. Angiotensin II blockers in obstructive pulmonary disease: a randomised controlled trial. Eur Respir J. 2006 May;27(5):972-9. doi: 10.1183/09031936.06.00098105. Epub 2006 Jan 30. PMID 16446313